CLINICAL TRIAL: NCT03402594
Title: Effects of High Flow Oxygen Therapy on Oxygen Desaturation Index in Patients With Acute Ischemic Stroke
Brief Title: High Flow Oxygen Therapy and Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 436/59
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-11

CONDITIONS: Stroke
Keywords: High flow oxygen therapy; Oxygen desaturation index; Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No oxygen (No Intervention): No oxygen supplementation given
- Low flow oxygen (Active Comparator): Oxygen cannula with a flow rate of 2 liter/minute
  Interventions: Device: Low flow oxygen
- High flow oxygen (Experimental): Heated humidified high flow oxygen cannula (Optiflow; temperature of 34°C and fractional inspired oxygen of 0.24) with a flow rate of 20 liter/minute
  Interventions: Device: High flow oxygen

INTERVENTIONS:
Device: High flow oxygen — Heated humidified high flow oxygen cannula (Optiflow; temperature of 34°C and fractional inspired oxygen of 0.24) with a flow rate of 20 liter/minute
  Arms: High flow oxygen
Device: Low flow oxygen — Oxygen cannula with a flow rate of 2 liter/minute
  Arms: Low flow oxygen

SUMMARY:
Hypoxemia is common in acute ischemic stroke and associated with neurological deterioration and mortality. However, the benefit of oxygen therapy is controversial. Severity of stroke may affect the benefit of oxygen supplementation. Abnormal breathing patterns are commonly found among stroke patients and may increase the risk of hypoxemia. High flow nasal cannula (HFNC) has several advantages from controllable fraction of inspired oxygen (FiO2), reduction of nasopharyngeal resistance and positive end expiratory pressure effect. In this study, we aimed to assess the therapeutic effect of HFNC on oxygen desaturation index (ODI) and neurological outcomes in stroke patients with moderate and severe severities, compared with no and low flow oxygen supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 or more
2. Clinical and radiographic findings including computerized tomography of brain compatible with acute ischemic stroke
3. Presentation within 72 hours after the stroke onset
4. National of Health Stroke Scale (NIHSS) of 5 or more,
5. Limb weakness defined as motor power grade of 4 or less,
6. Able to give informed consent, or the next of kin was willing to give assent

Exclusion Criteria:

1. Recognized indications for oxygen treatment, such as oxygen saturation on room air of less than 92%, acute left ventricular failure, severe pneumonia, pulmonary emboli, and chronic respiratory failure treated with home oxygen supplementation
2. Recognized contraindications for oxygen treatment including chronic hypercapnia and type II respiratory failure
3. Subjects with previous diagnosis of obstructive sleep apnea (OSA) or highly suspicious of OSA, screened by STOPBANG score of 5 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Oxygen desaturation index | In the first 24 hours of study period
  The number of times per hour that the oxygen saturation measured by pulse oximetry drop from baseline more than 4% for at least 10 seconds

SECONDARY OUTCOMES:
Mean oxygen saturation | In the first 24 hours of study period
Lowest oxygen saturation | In the first 24 hours of study period
The number of subjects with oxygen desaturation | In the first 24 hours of study period
Percentages of cumulative time of oxygen desaturation | In the first 24 hours of study period
NIHSS changes | at the 7th day of admission or at discharge date
  The NIHSS at randomization minus the NIHSS at the 7th day of admission
The number of subjects with NIHSS improvement by 4 or more | at the 7th day of admission or at discharge date